CLINICAL TRIAL: NCT03198806
Title: Influence of Hydration on Autonomic Behavior and Cardiorespiratory Parameters of Coronaropathy Submitted to Aerobic Exercise
Brief Title: Water Intake Associated With Aerobic Exercise in Coronary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Luiz Carlos Marques Vanderlei, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 54864716800005402
Record Dates: First submitted 2017-06-19; First posted 2017-06-26 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease
Keywords: Autonomic Nervous System; Fluid Therapy; Heart Rate; Exercise
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity | interventions — Supine Position; Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group in supine position (Active Comparator): Intervention:
  - Only treadmill aerobic exercise with 60 min recovery in supine position
  Interventions: Other: Treadmill aerobic exercise in supine position
- Hydration group in supine position (Experimental): Interventions:
  * Treadmill aerobic exercise with 60 min recovery in supine position
  * Water intake
  Interventions: Other: Treadmill aerobic exercise and water intake in supine position
- Control group in orthostatic position (Active Comparator): Intervention:
  - Only treadmill aerobic exercise with 10 min recovery in orthostatic position
  Interventions: Other: Treadmill aerobic exercise in orthostatic position
- Hydration group in orthostatic position (Experimental): Interventions:
  * Treadmill aerobic exercise with 10 min recovery in orthostatic position
  * Water intake
  Interventions: Other: Treadmill aerobic exercise and water intake in orthostatic position

INTERVENTIONS:
Other: Treadmill aerobic exercise in supine position — The volunteers will be submitted to a cardiovascular rehabilitation session with 40 minutes of treadmill aerobic exercise followed by 60 minutes of recovery at the supine position.
  Arms: Control group in supine position
Other: Treadmill aerobic exercise and water intake in supine position — The volunteers will be submitted to a cardiovascular rehabilitation session with 40 minutes of treadmill aerobic exercise and water intake followed by 60 minutes of recovery at the supine position.
  Arms: Hydration group in supine position
Other: Treadmill aerobic exercise in orthostatic position — The volunteers will be submitted to a cardiovascular rehabilitation session with 40 minutes of treadmill aerobic exercise followed by 10 minutes of recovery at the orthostatic position.
  Arms: Control group in orthostatic position
Other: Treadmill aerobic exercise and water intake in orthostatic position — The volunteers will be submitted to a cardiovascular rehabilitation session with 40 minutes of treadmill aerobic exercise and water intake followed by 10 minutes of recovery at the orthostatic position.
  Arms: Hydration group in orthostatic position

SUMMARY:
The need to restore water losses resulting from physical activity has become established and diffused into international consensus for healthy individuals or high-performance athletes. However, the influence of fluid replacement when administered during and after exercise on cardiorespiratory parameters, cardiac autonomic modulation, and subjective perceptions of effort and pain of individuals with autonomic alterations known as the coronary arteries remain poorly understood. In this sense, this study intends to investigate the influence of hydration on cardiac autonomic modulation, cardiorespiratory parameters, subjective perception of exertion and pain of coronary arteries submitted to aerobic exercise in the model of a cardiovascular rehabilitation session. A total of 31 individuals will be recruited in this study and will perform four standardized cardiovascular rehabilitation sessions. Only in the second and the fourth session will the volunteers be instructed to ingest a quantity of water predetermined by the evaluator, based on the loss of body mass measured in the first and the third sessions. The outcomes (autonomic modulation, cardiorespiratory variables and perceptions) will be evaluated before, during and after exercise. The results of this study will enable professionals working with this population to implement awareness strategies on the importance of fluid intake in cardiovascular rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Men with coronary heart disease ischemia, over 45 years
* At least three months of cardiovascular rehabilitation

Exclusion Criteria:

* smokers, alcoholics
* Uncontrolled metabolic disease (eg, uncontrolled diabetes and thyroid diseases)
* Abnormal hemodynamic responses during exercise such as disproportionate increase / fall of heart rate and / or blood pressure to low / high levels of load
* myocardial ischemia and / or severe ventricular arrhythmias during the exercise test

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | up to six months
  Indices of heart rate variability

SECONDARY OUTCOMES:
Subjective Effort Perception | up to six months
  Borg Scale
Subjective Pain Perception | up to six months
  Borg CR-10 Scale
Cardiovascular parameter | up to six months
  Heart Rate
Cardiovascular parameter | up to six months
  Blood Pressure
Cardiorespiratory parameter | up to six months
  Respiratory frequency
Cardiorespiratory parameter | up to six months
  Partial Oxygen Saturation

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Carlos Marques Vanderlei, PhD, Study Director — Universidade Estadual Paulista - UNESP - Campus de Presidente Prudente
Locations (1):
- Luiz Carlos Marques Vanderlei, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided